CLINICAL TRIAL: NCT06826066
Title: Involvement of the Immune System in Intrinsic Radiosensitivity
Acronym: TRANSPROUST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240671
Record Dates: First submitted 2025-01-30; First posted 2025-02-13 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TRANSPROUST is a prospective, single-center cohort. (Experimental)
  Interventions: Other: Blood samples

INTERVENTIONS:
Other: Blood samples — We propose to include patients who have been treated with radiotherapy and did not experience severe radiation-induced toxicity, after obtaining their informed consent. A blood sample will then be collected by the nursing staff from the Oncology-Radiotherapy department at Henri Mondor University Hospital. After the patient signs the consent form, each patient will have their clinical information recorded and a blood sample taken. The blood samples will be immediately transported, at room temperature, to the INSERM U955 i-Biot unit at Henri Mondor (serum, plasma, and PBMC). All samples will be frozen at -80°C for later analysis.

SUMMARY:
Radiotherapy is one of the major treatments for cancer. It may be indicated in more than two-thirds of patients, regardless of cancer location or disease stage. The mechanisms of radiotherapy action are numerous: halting tumor proliferation, inducing tumor cell death, triggering anti-tumor immune responses, and ensuring both local and systemic tumor control. As a result, current treatments are highly effective, providing, for instance, a 5-year overall survival rate of about 90%-95% for localized breast and prostate cancers.

DETAILED DESCRIPTION:
In everyday clinical practice, the indications for radiotherapy are based on the benefit-to-risk ratio concerning toxicity. In most cases, radiotherapy causes mild to moderate acute or late side effects, depending on the patient and the volumes irradiated. However, in 1% to 5% of treated patients, these side effects can be severe, unexpected, and often unexplained. The cause of this toxicity remains poorly understood and largely unexplored, especially concerning the intrinsic radiosensitivity of patients.

The PROUST study (French Registry for Review of Morbidity and Mortality; RMM) was initiated in France to prospectively collect clinical, dosimetric, and biological data on individual radiosensitivity in patients who experience severe radiation-induced toxicity. The goal of this study is to better characterize patients with severe radiation-induced toxicities and identify the cellular factors involved in this toxicity.

Although the aim is to identify the cellular and molecular immune factors involved in severe radiation-induced toxicity, we currently cannot determine whether the immune monitoring observed in radiosensitive patients is a consequence of the toxicity itself or of radiotherapy. To answer this question, we have decided to create a control cohort, called TRANSPROUST, which includes patients treated with radiotherapy but who did not experience severe radiation-induced toxicity. After obtaining consent from patients who were treated with radiotherapy but did not develop severe toxicity, we will collect blood samples similar to those taken from the severe toxicity cohort.

These samples will undergo flow cytometry analysis, and the results will be compared with those of patients included in the PROUST cohort.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients who have been treated with radiotherapy
* Absence of toxicity grade 2 or higher
* Patients without psychiatric, sociological, family, or geographical difficulties that could interfere with patient compliance to the protocol or follow-up
* Information and signed informed consent
* Affiliated with social security

Exclusion Criteria:

* Inability to obtain patient consent
* Patient refusing blood sample collection
* Patient deprived of liberty or under legal protection (under guardianship, under curatorship)
* Patients who have experienced radiation-induced toxicity of grade 2 or higher
* Disease progression, relapse
* Patient under State Medical Aid

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05-12 (Estimated); Study Completion 2027-05-12 (Estimated)

PRIMARY OUTCOMES:
Identify immunological markers predictive of intrinsic radiosensitivity. | 48 hours
  Identification of immunological markers predictive of intrinsic radiosensitivity using flow cytometry analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Henri Mondor, 1 rue Gustave Eiffel,, Créteil, Île-de-France Region, France

IPD SHARING:
Plan to Share IPD: No
DATA IS OWNED BY ASSISTANCE PUBLIQUE - HÔPITAUX DE PARIS